CLINICAL TRIAL: NCT00779948
Title: Dynamic Internal Fixation of Femoral Neck Fractures
Acronym: DIFINE
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-0806
Record Dates: First submitted 2008-10-16; First posted 2008-10-24 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Femoral Neck Fracture
Keywords: Femoral Neck Fracture; Internal Fixation; Dynamic Hip Screw
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Targon FN
- DHS

SUMMARY:
Evaluation of dynamic Plate-Screw-Systems for internal fixation after femoral neck fractures. Open Registry for Comparison of 1-screw-systems (DHS) with multi-screw-system Targon FN.

DETAILED DESCRIPTION:
Two implant systems are mainly used for internal fixation: canulated screws and plate-screw-systems. Regarding the latter, the dynamic hip screw systems (DHS)represent the most frequently used devices.

Targon FN (Aesculap) is a new plate-screw system and available on the market since 2007. In contrast to the DHS, which uses only one telescrew, the Targon FN provides up to four telescrews.

With this registry, we want to evaluate the results of Targon FN compared with DHS systems.

ELIGIBILITY:
Inclusion Criteria:

* men >= 60 years, women >= 55 years
* femoral neck fractures needing surgical therapy
* femoral head preserving indication
* Living in a 100 km Radius from Hospital

Exclusion Criteria:

* Patient not able to walk
* Previous fracture or surgery on ipsilateral hip
* pathological fracture
* open fracture

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Patients
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2008-12; Primary Completion 2012-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cumulative Complication Rate | 1 year

SECONDARY OUTCOMES:
Course of Surgery Mobilization Radiology functional Results (SF-12, IOWA Hip Score) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Helwig, Dr., Study Chair — University Hospital Freiburg
Locations (9):
- Germany (9):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Berufsgenossenschaftliche Klinik, Tübingen, Baden-Wurttemberg
  - Klinikum Bad Hersfeld GmbH, Bad Hersfeld, Hesse
  - Evangelisches Krankenhaus, Castrop-Rauxel, North Rhine-Westphalia
  - Raphaelsklinik, Münster, North Rhine-Westphalia
  - Marienkrankenhaus Schwerte gGmbH, Schwerte, North Rhine-Westphalia
  - Erzgebirgsklinikum Annaberg gGmbH, Annaberg-Buchholz, Saxony
  - Krankenhaus Bethel, Berlin, State of Berlin
  - BGU Ludwigshafen, Ludwigshafen